CLINICAL TRIAL: NCT05779280
Title: Prospective, Double-Blinded, Randomized Head-to-Head Study of Topical Acetyl Zingerone With Teterahexyldecyl Ascorbate (THDA) Versus THDA Alone
Brief Title: Prospective Study of Topical Vitamin C (THDA) Versus Topical Vitamin C (THDA) With Acetyl Zingerone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Sytheon Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOP_AZ_THDA
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Wrinkle; Skin Pigmentation
Keywords: Vitamin C; Acetyl Zingerone
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THDA + Acetyl Zingerone (Experimental): Product will be used twice daily- once in the morning and once in the evening for 8 weeks. Each application will consist of 1-2 pumps (size of quarter) onto the face and neck, until fully absorbed.
  Interventions: Other: THDA + Acetyl Zingerone Topical Product
- THDA only (Active Comparator): Product will be used twice daily- once in the morning and once in the evening for 8 weeks. Each application will consist of 1-2 pumps (size of quarter) onto the face and neck, until fully absorbed.
  Interventions: Other: THDA

INTERVENTIONS:
Other: THDA + Acetyl Zingerone Topical Product — A skin care product with Acetyl Zingerone (Synoxyl® AZ) and THDA (VitaSynol® C) used twice daily
  Arms: THDA + Acetyl Zingerone
Other: THDA — A skin care product with THDA (VitaSynol® C) used twice daily
  Arms: THDA only

SUMMARY:
The purpose of this study is to asses the impact of topically applying a form of vitamin C known as tetrahexyldecyl Ascorbate (THDA) along with a novel anti-aging ingredient, acetyl zingerone, compared against applying THDA alone.

DETAILED DESCRIPTION:
In this study, we examine the effects of adding acetyl zingerone to vitamin-C derived ester THDA on its effects on the signs of photoaging (redness, uneven skin tone, and the appearance of fine lines) and compare it to the effects of applying THDA alone.

Acetyl zingerone is derived from ginger and has anti-oxidant properties

In this study, participants will be randomized to either receiving a THDA + acetyl zingerone product or a THDA only product.

This means that you will have an equal chance of receiving either product. You and the research team will not know which product you have been randomized to received because the products will be labelled with a code. The research team will only know which product contained THDA + acetyl zingerone and which product contained only THDA at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 30 years old and 65 years old.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Subjects using any topical retinoid, acetyl zingerone, vitamin C, bakuchiol, hyaluronic acid or benzoyl peroxide containing topical product within 2 weeks of starting study or any subject unwilling to refrain from washout prior to enrollment.
* Subjects with any of the following facial cosmetic treatments in the past 3 months or those who are unwilling to withhold the following facial cosmetic treatments during study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Facial fine lines and wrinkles | 8 weeks
  Change in severity of fine lines and wrinkles measured by photographic analysis (BTBP 3D Camera System)
Facial skin pigment evenness | 8 weeks
  Change in the appearance of facial skin pigment intensity measured by photographic analysis (BTBP 3D Camera System)

SECONDARY OUTCOMES:
Facial fine lines and wrinkles | 4 weeks
  Change in severity of fine lines and wrinkles measured by photographic analysis (BTBP 3D Camera System)
Facial skin pigment evenness | 4 weeks
  Change in the appearance of facial skin pigment intensity measured by photographic analysis (BTBP 3D Camera System)
Skin redness | 4 weeks
  Change in the appearance of skin redness measured by photographic analysis (BTBP 3D Camera System)
Skin redness | 8 weeks
  Change in the appearance of skin redness measured by photographic analysis (BTBP 3D Camera System)
Change in skin pigmentation in the undereye area | 4 weeks
  hange in skin pigmentation in the undereye area by Skin colorimetric analysis of pigment
Change in skin pigmentation in the undereye area | 8 weeks
  hange in skin pigmentation in the undereye area by Skin colorimetric analysis of pigment
Self-perception of skin parameters | 4 weeks
  Survey based self-assessment of facial features such as fine lines and wrinkles, skin smoothness, skin firmness
Self-perception of skin parameters | 8 weeks
  Survey based self-assessment of facial features such as fine lines and wrinkles, skin smoothness, skin firmness
Tolerability of product | 4 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin product
Tolerability of product | 8 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin product

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No